CLINICAL TRIAL: NCT05572619
Title: An Open Label, Single-center, Retrospective, Pivotal Study to Evaluate the Efficacy of Clinical Decision Support System for Large Vessel Occlusion Using Brain CT Images
Brief Title: Evaluation of Clinical Decision Support System for Large Vessel Occlusion Using Brain CT Images
Status: Completed | Type: Observational
Sponsor: Heuron Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HR-cELVO-01
Record Dates: First submitted 2022-10-04; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Norwood Procedures; Fontan Procedure

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 14 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive group: A patient diagnosed with large vessel occlusion after a non-contrast CT, CT perfusion and CT angiography
  Interventions: Device: 1st Reading; Device: 2nd Reading
- Negative group: A normal person or a patient not diagnosed with intracranial haemorrhage after a non-contrast CT, CT perfusion and CT angiography
  Interventions: Device: 1st Reading; Device: 2nd Reading

INTERVENTIONS:
Device: 1st Reading — The medical team visually checks the non-contrast CT without cELVO and diagnose the large vessel occlusion.
  Other Names: Stage 1
Device: 2nd Reading — The medical team visually checks the non-contrast CT with assistance from the cELVO and diagnose the large vessel occlusion.
  Other Names: Stage 2

SUMMARY:
cELVO is a software that has been pre-learned based on a large vessel occlusion diagnosis model using brain CT images, and clinical decision support system for diagnosing large vessel occlusion by automatically analyzing brain CT images by assisting the medical team.

The specific aims of this study are to evaluate efficacy of cELVO compared to the sensitivity and specificity levels of medical team to diagnosis with and without cELVO used.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 19 years old
* Brain non-contrast CT, CT perfusion and CT angiography acquired
* Positive group: A patient diagnosed with large vessel occlusion after a non-contrast CT, CT perfusion and CT angiography
* Negative group: A normal person or a patient not diagnosed with large vessel occlusion after a non-contrast CT, CT perfusion and CT angiography

Exclusion Criteria:

* Poor or incomplete brain non-contrast CT, CT perfusion and CT angiography quality

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (1) Adults over 19 years old (2) Brain non-contrast CT, CT perfusion and CT angiography acquired (3) who confirmed with large vessel occlusion(positive group) or not large vessel occlusion or normal(negative group)
Sampling Method: Probability Sample
Enrollment: 479 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of medical team compared with/without cELVO | Within 2 weeks after completion of reading
  Sensitivity and specificity of determining large vessel occlusion of medical team when using cELVO compared to not using cELVO

SECONDARY OUTCOMES:
Accuracy of medical team compared with/without cELVO | Within 2 weeks after completion of reading
  Accuracy of determining large vessel occlusion of medical team when using cELVO compared to not using cELVO
ROC Curve for medical team compared with/without cELVO | Within 2 weeks after completion of reading
  ROC Curve of determining large vessel occlusion of medical team when using cELVO compared to not using cELVO
AUC values for medical team compared with/without cELVO | Within 2 weeks after completion of reading
  AUC values of determining large vessel occlusion of medical team when using cELVO compared to not using cELVO
Sensitivity and specificity of each reader compared with/without cELVO | Within 2 weeks after completion of reading
  Sensitivity and specificity of determining large vessel occlusion of each reader when using cELVO compared to not using cELVO
Sensitivity and specificity of cELVO | Within 2 weeks after completion of reading
  Sensitivity and specificity of cELVO in diagnosis of large vessel occlusion based on golden standards

CONTACTS AND LOCATIONS:
Overall Officials: Myeong Jin Kim, M.D.pH.D, Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Gachon University Gil Medical Center, Incheon, Namdong-gu, South Korea

IPD SHARING:
Plan to Share IPD: No